CLINICAL TRIAL: NCT01269879
Title: Vibration Training in Epicondylitis - a Randomized Trial
Brief Title: VIBration Training in EpicondylitiS
Acronym: VIBES
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Hannover Medical School, Karsten Knobloch, MD, PHD, FACS, Hannover Medical School, Plastic, Hand and Reconstructive Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIBES-2010
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Epicondylitis; Pain; Tendinopathy
Keywords: epicondylitis; pain; tendon
MeSH Terms: conditions — Pain; Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active control (Flexi-Bar only) (Active Comparator): Flexi-Bar vibration training only over 12 weeks with three distinct exercises and 10min training twice daily
  Interventions: Device: Flexi-Bar vibration device only
- Intervention Flexi-Bar + XCO-Trainer (Experimental): Combination intervention using vibration device Flexi-Bar and XCO-Trainer (oscillating mass witin a tube moved during running 40-60min/week suggested)
  Interventions: Device: Flexi-Bar + XCO-Trainer

INTERVENTIONS:
Device: Flexi-Bar vibration device only — daily vibration training 10min twice
  Other Names: vibration; Flexi bar
  Arms: Active control (Flexi-Bar only)
Device: Flexi-Bar + XCO-Trainer — XCO-Trainer is a way to overload the cardiovascular system and the core muscles during running. An oscillating mass inside the XCO-Trainer is activated when the XCO is propelled forward and backward with force. The movement of the mass triggers a series of responses from the runners' body.
  In addition Flexi-Bar vibration training as in the referred active comparator group
  Other Names: XCO; XCO Trainer; Flexibar; vibration
  Arms: Intervention Flexi-Bar + XCO-Trainer

SUMMARY:
A number of different therapeutic approaches to treat lateral epicondylitis have been tested partly in randomized trials, such as polidocanol sclerosing injections, botulinom toxin A injections, braces, surgery and topical NO patches.

One study indicates that patients with lateral epicondylitis (lateral elbow tendinopathy) have poorer elbow proprioception in contrast to healthy controls (Juul-Kristensen B, et al., J Shoulder Elbow Surg 2008;17(1 Suppl):72S-81S.)

Based on a suggested poorer elbow proprioception in lateral elbow tendinopathy, The investigators hypothesize that a dedicated proprioceptive intervention might be able to reduce pain and improve function.

As such a RCT is planned with two intervention arms with proprioceptive training using the Flexi-Bar vibration device (www.flexi-bar.co.uk) +/- the XCO-Trainer (www.xco-trainer.co.uk) over twelve weeks.

DETAILED DESCRIPTION:
The investigators sought to evaluate the clinical effects of either a vibration training using the Flexi-Bar vibration device (www.flexi-bar.co.uk) +/- the XCO-Trainer (www.xco-trainer.co.uk) in a randomized trial among patients suffering lateral elbow tendinopathy (lateral epicondylitis).

Primary outcome measure of this clinical trial is pain on a visual analogue scale (VAS 0-10) before and after 12 weeks of training.

Secondary outcome parameters involve DASH score before and after, grip strength (JAMAR), vibration and two-point discrimination (mm).

ELIGIBILITY:
Inclusion Criteria:

* lateral elbow tendinopathy
* informed consent
* ability to run at least 40-60min per week with a XCO-Trainer device

Exclusion Criteria:

* other sources of lateral elbow pain (joint instabilities, fractures)
* no consent
* no ability to run at least 40-60min per week using a XCO-Trainer device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Pain on a visual analogue scale (VAS 0-10) | before and 12 weeks after
  Pain on VAS (0=no pain at all, 10= worst pain imaginable) before and 12 weeks after the intervention.

SECONDARY OUTCOMES:
DASH Score | before and 12 weeks after
  DASH score (0=no impairment, 100=severe impairment) of daily activities
Grip strength (JAMAR) | before and after 12 weeks
  Grip strength (JAMAR) in two elbow positions (0° flexion, 90° flexion) before and after 12 weeks of intervention
Vibration | before and 12 weeks after
  Vibration using a 128Hz tuning fork before and 12 weeks after the intervention
2-point discrimination | before and 12 weeks after the intervention
  2-point discrimination (mm) before and after the intervention and the finger tips

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Knobloch, FACS, MD, PhD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Plastic, Hand and Reconstructive Surgery, Hanover, Germany

REFERENCES:
- [Background] Knobloch K. Lateral elbow tendinopathy. Am J Sports Med. 2010 Nov;38(11):NP3; author reply NP3-4. doi: 10.1177/0363546510383492. No abstract available. PMID 20971969
- [Background] Knobloch K. [Non-operative therapy in lateral epicondylitis]. MMW Fortschr Med. 2009 Feb 19;151(8):28-30. No abstract available. German. PMID 19432271
- [Background] Knobloch K. Re: Radiofrequency microtenotomy: a promising method for treatment of recalcitrant lateral epicondylitis. Am J Sports Med. 2008 Nov;36(11):e2-3; author reply e3. doi: 10.1177/0363546508325661. No abstract available. PMID 18978181
- [Background] Knobloch K, Spies M, Busch KH, Vogt PM. Sclerosing therapy and eccentric training in flexor carpi radialis tendinopathy in a tennis player. Br J Sports Med. 2007 Dec;41(12):920-1. doi: 10.1136/bjsm.2007.036558. Epub 2007 May 11. PMID 17496066
- [Background] Knobloch K. [Eccentric exercise in tendinopathies]. Sportverletz Sportschaden. 2010 Dec;24(4):187. doi: 10.1055/s-0029-1245845. Epub 2010 Dec 14. No abstract available. German. PMID 21157652
- [Background] Knobloch K, Gohritz A. Dr Runge: a German pioneer in sclerosing therapy in epicondylitis in 1873. Br J Sports Med. 2010 Nov 16. doi: 10.1136/bjsm.2008.051326. Online ahead of print. No abstract available. PMID 21081643
- [Background] Yoon U, Knobloch K. Reporting quality in evidence-based studies. J Am Coll Surg. 2010 Apr;210(4):533. doi: 10.1016/j.jamcollsurg.2009.12.028. No abstract available. PMID 20347748
- [Background] Yoon U, Knobloch K. Quality of reporting in sports injury prevention abstracts according to the CONSORT and STROBE criteria: an analysis of the World Congress of Sports Injury Prevention in 2005 and 2008. Br J Sports Med. 2012 Mar;46(3):202-6. doi: 10.1136/bjsm.2008.053876. Epub 2009 Jul 26. PMID 19656768
- [Background] Juul-Kristensen B, Lund H, Hansen K, Christensen H, Danneskiold-Samsoe B, Bliddal H. Poorer elbow proprioception in patients with lateral epicondylitis than in healthy controls: a cross-sectional study. J Shoulder Elbow Surg. 2008 Jan-Feb;17(1 Suppl):72S-81S. doi: 10.1016/j.jse.2007.07.003. Epub 2007 Nov 26. PMID 18036844
- [Background] Garg R, Adamson GJ, Dawson PA, Shankwiler JA, Pink MM. A prospective randomized study comparing a forearm strap brace versus a wrist splint for the treatment of lateral epicondylitis. J Shoulder Elbow Surg. 2010 Jun;19(4):508-12. doi: 10.1016/j.jse.2009.12.015. Epub 2010 Apr 2. PMID 20363158
- [Background] Mileva KN, Kadr M, Amin N, Bowtell JL. Acute effects of Flexi-bar vs. Sham-bar exercise on muscle electromyography activity and performance. J Strength Cond Res. 2010 Mar;24(3):737-48. doi: 10.1519/JSC.0b013e3181c7c2d8. PMID 20145560